CLINICAL TRIAL: NCT04533841
Title: Propranolol and Misoprostol Versus Misoprostol Alone for Induction of Labor In Primigravidas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ahmed mohamed fathy ismail (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Sponsor-Investigator, Ahmed mohamed fathy ismail, Director, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ahmed mohamed fathy ismail
Record Dates: First submitted 2020-08-26; First posted 2020-09-01 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Induction of Labor Affected Fetus / Newborn
MeSH Terms: interventions — Misoprostol; Propranolol

STUDY DESIGN:
Intervention Model Description: Clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded research
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Misoprostol + propranolol (Active Comparator): Patient who receive misoprostol then after 30minutes receive propranolol
  Interventions: Drug: Misoprostol; Drug: Propranolol
- Misoprostol + placebo (Placebo Comparator): Pt who will receive misoprostol then after 30minutes receive placebo
  Interventions: Drug: Misoprostol; Drug: Placebo

INTERVENTIONS:
Drug: Misoprostol — Pt will receive misoprostol for labor induction then after 30 minutes will receive ether propranolol or misoprostol
Drug: Placebo — placebo
  Arms: Misoprostol + placebo
Drug: Propranolol — Propranolol
  Arms: Misoprostol + propranolol

SUMMARY:
To compare propranolol and misoprostol versus misoprostol alone for induction of labour in primigravidas

DETAILED DESCRIPTION:
Candidates will be randomized into 2 groups according to a computer generated sequence. Each candidate will be assigned an opaque sealed envelope containing a paper with her group on it. Both the patient and doctor on duty will be blinded to which group the patient was assigned to.

- Study procedure:

1. Written informed consent will be obtained from all participants prior to the study.
2. Full history taking.
3. General examination.

Patients will be subjected to the following:

* Patients attending labour room for induction of labour will be divided into two groups.
* Both groups, women are induced with Tab misoprostol 25μg applied to posterior vaginal fornix under aseptic precaution and every 6 hours for a maximum of 4 doses.
* In group 1, after induction is started with misoprostol placement, 30 minutes will pass before administration of oral Propanolol 20mg
* In group 2, after induction is started with misoprostol placement, 30 minutes will pass before administration of oral placebo in the form of sugary tablets.
* After induction, women will be monitored for fetal and maternal wellbeing and progress of labour.

ELIGIBILITY:
Inclusion Criteria:

* • Primigravidas.

  * Full term patients with ultrasound confirmed dates.
  * Singleton.
  * Cephalic presentation.
  * Fetal heart rate between 120 to 160 beats per minute.

Exclusion Criteria:

* • Any history of previous surgery on the uterus.

  * Patients in active labour, with ruptured membranes.
  * Fetal distress.
  * Macrosomia or polyhydramnios
  * Hypersensitivity to prostaglandins.
  * Asthmatic patient .
  * liver or kidney impairment .
  * known cardiac patient with abnormal ECG.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female full term pregnancy primigravida
Enrollment: 128 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-09-13 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Induction delivery interval | procedure delivery
  The time from starting induction to the delivery

SECONDARY OUTCOMES:
Mode of delivery | delivery
  Vaginal delivery or cesarian section

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed S Abd El hamid, A.professor, Study Director — Ain Shams University; Hazem A Hassan elzeneiny, Professor, Study Director — Ain Shams University
Locations (1):
- Ahmed mohamed fathy ismail, Zagazig, El Sharquia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study results will be available
Supporting Information: Study Protocol, CSR
Time Frame: September 2020
Access Criteria: Researchers

REFERENCES:
- [Derived] Abdel Hamid AS, El Zeneiny H, Fathy A, Nawara M. A pilot study to compare propranolol and misoprostol versus misoprostol and placebo for induction of labor in primigravidae; a randomized, single-blinded, placebo-controlled trial. BMC Pregnancy Childbirth. 2023 Apr 4;23(1):226. doi: 10.1186/s12884-023-05537-1. PMID 37016326